CLINICAL TRIAL: NCT07261488
Title: The Impact of Inaccurate Wound Assessment on Treatment Efficiency: A Multicenter Cross-Sectional Survey in the Beijing-Tianjin-Hebei Region of China
Brief Title: Wound Assessment Accuracy and Treatment Efficiency
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Head of Wound Healing Center, Peking University Third Hospital
Other Study IDs: Long2025-WC-wound assessment
Record Dates: First submitted 2025-10-01; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Wound - in Medical Care
Keywords: Wound Assessment; Wound healing; Accuracy; Efficacy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- wound care group: It involved 118 wound specialists from 9 specialized wound care institutions in the Beijing-Tianjin-Hebei region of China

SUMMARY:
Wound assessment is critical for developing effective treatment strategies, yet there is a scarcity of research on the assessment accuracy of clinical practitioners. An online questionnaire-based survey was conducted from March to April 2025. It involved 118 wound specialists from 9 specialized wound care institutions in the Beijing-Tianjin-Hebei region of China, who evaluated 8 standardized wound cases. A total of 553 valid responses were collected.

ELIGIBILITY:
Inclusion Criteria:

* being a wound therapist, specialized nurse, or physician in relevant departments;
* having completed systematic specialized wound training (provided by, but not limited to, EWMA, ICW, ET, the Chinese Nursing Association, the Wound Baihui online education platform, or other medical institutions)

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 553 valid responses were collected
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
The weighted overall accuracy of wound assessments | Baseline
  Compare the assessment answers given by wound specialist to determine the accuracy rate of the assessment of the wound practitioners surveyed

SECONDARY OUTCOMES:
The average accuracy for observational assessment items (e.g., wound size, types of wound bed tissue, wound exudate) | Baseline
  An assessment response was scored as correct if it was consistent with the standard answer. Calculate the accuracy for observational assessment items (e.g., wound size, types of wound bed tissue, wound exudate) .
The average the accuracy of inferential assessment items (e.g., etiologic classification of wounds, healing capacity, wound characteristic analysis) | Baseline
  An assessment response was scored as correct if it was consistent with the standard answer. Calculated the average accuracy of inferential assessment items (e.g., etiologic classification of wounds, healing capacity, wound characteristic analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Samaniego-Ruiz MJ, Llatas FP, Jimenez OS. Assessment of chronic wounds in adults: an integrative review. Rev Esc Enferm USP. 2018 Jun 25;52:e03315. doi: 10.1590/S1980-220X2016050903315. English, Spanish. PMID 29947700
- [Result] Koschwanez HE, Broadbent E. The use of wound healing assessment methods in psychological studies: a review and recommendations. Br J Health Psychol. 2011 Feb;16(Pt 1):1-32. doi: 10.1348/135910710X524633. PMID 21226781